CLINICAL TRIAL: NCT06251609
Title: Naloxone for Opioid Associated Out of Hospital Cardiac Arrest
Acronym: NOPACA
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NOPACAV1
Record Dates: First submitted 2024-01-19; First posted 2024-02-09 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Heart Arrest, Out-Of-Hospital; Opioid Overdose; Naloxone
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Opiate Overdose | interventions — Naloxone; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Naloxone (Active Comparator): The intervention consists of naloxone 2mg (2ml of 1mg/ml solution) administered by EMS personnel via the IV or IO route. The study intervention will be administered immediately (within 5 minutes) following the first dose of epinephrine.
  Interventions: Drug: Naloxone 2 MG
- Saline (Placebo Comparator): Saline 2ml will be supplied in pre-filled syringes within numbered trial treatment packs. The trial will be double-blind; patients, investigators, and the clinical team will be blinded. Only the pharmacy providing the numbered syringes will be aware of the allocation but will not be involved with clinical care or outcome evaluation. The saline placebo will be stored in syringes identical to the naloxone syringes without identifying features.
  Interventions: Drug: Saline 2ml

INTERVENTIONS:
Drug: Naloxone 2 MG — The intervention consists of naloxone 2mg (2ml of 1mg/ml solution) administered by EMS personnel via the IV or IO route. The study intervention will be administered immediately (within 5 minutes) following the first dose of epinephrine. When naloxone hydrochloride is administered intravenously, the onset of action is generally apparent within two minutes. The naloxone will be administered following the first dose of epinephrine. The control is saline 2ml will be supplied in pre-filled syringes within numbered trial treatment packs. They will be identical in appearance to the naloxone syringes.
  Other Names: narcan
  Arms: Naloxone
Drug: Saline 2ml — Placebo
  Arms: Saline

SUMMARY:
The investigator's long-term goal is to conduct Naloxone for Opioid Associated out of Hospital Cardiac Arrest (NOPACA), a randomized, double blind, controlled trial to determine the efficacy of naloxone vs. placebo in Opioid Associated out of Hospital Cardiac Arrest. The investigative team plan to randomize patients in OHCA to early naloxone administration vs. placebo after initial resuscitation and measure ROSC and survival. Challenges to designing NOPACA include uncertainty regarding: 1) the available pool of participants and number of EMS agencies needed to meet enrollment targets; 2) acceptability among patients, EMS and Emergency Medicine provider stakeholders, and 3) estimates of the study outcomes needed for sample size estimates. Toward obtaining the necessary information to design NOPACA, the investigators propose a pilot RCT of participants at high risk for OA-OHCA to verify a reasonable recruitment rate; treatment fidelity and acceptability; and adequate retention and measurement of outcomes at follow up. The investigators propose incorporating hypothesis testing of the feasibility outcomes to determine progression to a definitive trial.

DETAILED DESCRIPTION:
Rationale: Opioid associated out-of-hospital cardiac arrest (OA-OHCA) is defined as cardiac arrest precipitated by the use of opioids, with or without co-intoxicants and comorbidities. In OA-OHCA, hypoxia is thought reduce cardiac output, resulting in hypotension, bradycardia, and pulseless electric activity (PEA) or asystole. This pathophysiology is distinct from sudden cardiac death and other arrest etiologies and may benefit from targeted treatments, including naloxone. Naloxone is a competitive mu opioid-receptor antagonist that reverses the central nervous system, respiratory, and circulatory effects of opioids. Naloxone improves cardiac arrest outcomes in animals, and a recent retrospective analysis of cardiac arrests from 1300 EMS agencies found that survival and return of spontaneous circulation (ROSC) were higher in those given naloxone compared to those not receiving naloxone in patients presenting in PEA. Whether naloxone benefits patients in OA-OHCA is a knowledge gap that should be assessed in a randomized controlled trial.

The long-term goal is to conduct Naloxone for Opioid Associated Out of Hospital Cardiac Arrest (NOPACA), a randomized, controlled trial to determine the efficacy of naloxone vs. placebo in OA-OHCA. To design NOPACA, the investigators propose a pilot RCT of participants at high risk for OA-OHCA to verify a reasonable recruitment rate; treatment fidelity; and adequate retention and measurement of outcomes at follow up.

Hypothesis: The overall hypothesis is that early EMS administration of naloxone (in addition to standard resuscitation) improves survival in patients in OA-OHCA. The hypothesis of the pilot RCT is that the investigators can feasibly enroll, randomize, administer naloxone, and measure ROSC and survival at hospital discharge.

Aim 1: Determine the ability to enroll and randomize participants into a RCT of naloxone vs. placebo for OA-OHCA.

Aim 2: Determine the ability to deliver the treatments per protocol, after standard initial resuscitation measures (within 5 minutes of initiating CPR and giving the first dose of epinephrine).

Aim 3: Determine the ability to measure primary efficacy outcomes (rate of ROSC at ED arrival and survival at hospital discharge)23 and obtain a preliminary estimate of effect size for the future trial.

Design: Pilot, randomized, parallel group, placebo-controlled trial. Study population: Participants are adults in EMS attended out of hospital cardiac arrest, in whom EMS has initiated ACLS treatment, including ventilation, CPR, and obtain IV/IO access and administered epinephrine. Based on prior research to identify patients at high risk of OA-OHCA, participants meeting less than 60 years old who receive initial resuscitation measures will be eligible for inclusion.

Setting: The University of California, San Francisco and San Francisco Fire Department Fire Department.

Intervention: Naloxone 2mg (2ml of 1mg/ml solution) administered by EMS personnel via the IV (or IO) route immediately (within 5 minutes) following the first dose of epinephrine.

Control: Saline 2ml will be supplied in pre-filled syringes within numbered trial treatment packs.

Feasibility outcomes will allow the investigators to determine whether the NOPACA future trial is feasible and estimate how many sites might be needed.

* Number of EMS treated OHCA patients who meet inclusion criteria per month, with a goal of > 3 per month
* Proportion of those randomized participants who receive the study drug based on randomization assignment, with a target treatment fidelity ≥ 75%.
* Proportion of randomized participants who are retained in the study, with a goal of retention and ascertainment of outcomes in ≥ 75% of participants.

Efficacy outcomes include sustained ROSC, survival to hospital discharge, and neurologic outcome will be assessed with the modified Rankin Scale.

Statistical analyses and reporting will adhere to CONSORT guidelines. The two groups will be compared in relation to baseline patient and cardiac arrest characteristics using descriptive statistics. All analyses of outcomes will be conducted on an intention-to-treat basis including patients randomized to a study arm and meeting all inclusion criteria and no known exclusion criteria at the time of drug administration. Point and confidence estimates will be the preferred measure to report group differences and all confidence intervals will have 95% coverage. All tests will be two-sided, and a p-value <0.05 will be considered significant Significance: By conducting Pilot-NOPACA, the investigators will determine whether the plan for NOPACA, a definitive trial of naloxone for OA-OHCA, is feasible. Also, the investigators will have obtained the regulatory approvals, including Exception from Informed Consent. Determining the benefit of naloxone in OA-OHCA is an American Heart Association research priority and may save thousands of lives each year in a worsening opioid epidemic.

ELIGIBILITY:
Inclusion Criteria:

Patients will be eligible if all the following criteria are met:

• Adults (age ≥ 18 years) in OHCA per EMS protocol. ACLS interventions have been initiated by EMS: chest compressions, ventilation; • 1st dose of epinephrine given via IV or IO.

•. At risk of OA-OHCA (EMS presumed drug-related OHCA or NACARDI positive for occult OA-OHCA) as described above.

Exclusion Criteria:

* EMS plans to administer naloxone, or administration of naloxone by EMS during the same encounter
* Cardiac arrest apparently caused by trauma, choking, or drowning.
* Known or apparent pregnancy
* Patient experiences ROSC prior to study drug administration
* Prior inclusion in the study
* Patient has an opt out bracelet or family member states exclusion •. Children less than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2026-11 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Survival to hospital discharge | Through hospital discharge, an average of up to 5 days
  Survival to hospital discharge is defined as patient is discharged from the hospital acute care unit alive regardless of neurological status, outcome or destination.

SECONDARY OUTCOMES:
Sustained Return of Spontaneous Circulation (ROSC) | Through completion of the index EMS encounter, an average of 30 minutes
  Palpable pulses or other signs of circulation without a need for chest compressions lasting at least 20 minutes or with pulse at time of transfer of care to the ED.

OTHER OUTCOMES:
Sufficient subjects to conduct the trial | Monthly, throughout duration of the trial
  Number of EMS treated OHCA patients who meet inclusion criteria per month
Proportion of OHCA eligible for study | Monthly, throughout duration of the trial
  Proportion of all EMS OHCA cases that meet all inclusion criteria and no exclusion criteria
Study Drug administration compliance | Between time of randomization and end of EMS encounter, an average of 30 minutes
  Proportion of those randomized participants who receive the study drug based on randomization assignment, with a target treatment fidelity ≥ 75%.
Participant retention | Through study completion and outcome ascertainment, and average of up to 5 days
  Proportion of randomized participants who are retained in the study, with a goal of retention and ascertainment of outcomes in ≥ 75% of participants.

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Wang, MD, MAS, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, Analytic Code